CLINICAL TRIAL: NCT04836767
Title: Evaluation of Exercise Capacity, Peripheral Muscle Strength, Balance, Cognitive Status and Quality of Life in Patients With COVID-19 in Long Term
Brief Title: Evaluation of Physical and Functional Status in Patients With COVID-19 in Long Term
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Associate Professor, Hacettepe University
Other Study IDs: GO21-178
Record Dates: First submitted 2021-04-07; First posted 2021-04-08 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Corona Virus Infection; Covid19
Keywords: COVID-19; SARS-CoV2; pandemic; post-COVID-19; exercise capacity
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- people with a history of COVID-19: COVID-19 Group Inclusion Criteria
  * Having been diagnosed with COVID-19 at least 12 weeks ago,
  * Being literate,
  * Being in the age range of 18-65,
  * Volunteering to participate in research,
  * To be clinically stable, to be under control if any accompanying comorbid conditions (such as hypertension, diabetes),
  * Not having any orthopedic and neurological problems that might interfere with evaluating peripheral muscle strength, balance and exercise capacity.
  COVID-19 Group Exclusion Criteria
  * Those with an ICU hospitalization history due to the diagnosis of COVID-19,
  * Recent myocardial infarction and pulmonary embolism.
  * Having accompanying chronic diseases,
  * Those who have any orthopedic or neurological disorders that will prevent walking,
  * Another COVID-19 PCR Test positivity in the last 12 weeks,
  * Not being able to cooperate and adapt to exercise test due to neurological influences such as cerebrovascular disease or psychiatric disorders,
- healthy people: Healthy Group Inclusion Criteria
  * Not having COVID-19,
  * Being literate,
  * Being in the age range of 18-65,
  * Volunteering to participate in research. The Criteria for Not Including the Healthy Group in the Study
  * Those who have any orthopedic or neuromuscular disorders that will prevent walking,
  * Having any chronic illness or psychiatric conditions or mental afflictions that may interfere with cooperation or compliance with exercise tests.

SUMMARY:
The reason the investigators want to do this research; Especially after Covid-19 infection, no research has been found on functional status in the long term. Therefore, in our study, the investigators aimed to evaluate exercise capacity, functional status, peripheral muscle strength, balance, anxiety and depression level, consciousness, work productivity, pain, fear of movement, and quality of life in patients with Covid-19 and to compare them with healthy individuals who have not had COVID-19.

DETAILED DESCRIPTION:
In our study, the investigators aimed to evaluate long-term exercise capacity, functional status, peripheral muscle strength, balance, anxiety and depression level, cognitive status, pain, kinesophobia and quality of life in patients with COVID-19, and to compare them with healthy individuals who have not had COVID-19. Our second goal; It is the evaluation of the relationship between long-term exercise capacity, pain, kinesiophobia, peripheral muscle strength, balance, anxiety and depression level, cognitive status and quality of life in individuals with COVID-19. It will also be examined whether these parameters change according to the post-COVID functional restriction level.

3. Materials and Methods of the Research: 3.1. The place of the study: Cardiopulmonary Rehabilitation Unit of Hacettepe University Faculty of Physical Therapy and Rehabilitation and Hacettepe University Faculty of Medicine Department of General Internal Medicine

3.2. Time of the study: It is planned to collect data and write the study between February 2021 and February 2022.

3.3. Research population, sample, research group:

The population of the study is individuals who have passed the diagnosis of COVID-19 for at least 12 weeks and healthy individuals who have not had COVID-19.

The sample of the study is individuals in the long-term after the diagnosis of COVID-19 at least 12 weeks after the diagnosis of COVID-19 in Hacettepe University Adult Hospital who meet the inclusion criteria and volunteer to participate in the study, and healthy individuals who have not had COVID-19.

Study Design:

Individuals meeting the inclusion criteria will be included in the study. The study will be conducted with people between the ages of 18-65, whose education level is at least primary school, and whose local language is Turkish. A total of 40 participants, 20 healthy without COVID-19, and 20 with at least 12 weeks past the diagnosis of COVID-19, will be included in the study. The guidance of the participants will be provided by the relevant physicians of the General Internal Medicine Unit of Hacettepe University Internal Diseases Department.

In accordance with the COVID-19 pandemic precautions, social distance rules will be followed in the tests to be carried out with individuals, care will be taken to use masks, and the materials to be used in tests and measurements will be disinfected before and after use.

COVID-19 Group Inclusion Criteria

* Having been diagnosed with COVID-19 at least 12 weeks ago,
* Being literate,
* Being in the age range of 18-65,
* Volunteering to participate in research,
* To be clinically stable, to be under control if any accompanying comorbid conditions (such as hypertension, diabetes),
* Not having any orthopedic and neurological problems that might interfere with evaluating peripheral muscle strength, balance and exercise capacity.

COVID-19 Group Exclusion Criteria

* Those with an ICU hospitalization history due to the diagnosis of COVID-19,
* Recent myocardial infarction and pulmonary embolism.
* Having accompanying chronic diseases,
* Those who have any orthopedic or neurological disorders that will prevent walking,
* Another COVID-19 PCR Test positivity in the last 12 weeks,
* Not being able to cooperate and adapt to exercise test due to neurological influences such as cerebrovascular disease or psychiatric disorders,

Healthy Group Inclusion Criteria

* Not having COVID-19,
* Being literate,
* Being in the age range of 18-65,
* Volunteering to participate in research.

The Criteria for Not Including the Healthy Group in the Study

* Those who have any orthopedic or neuromuscular disorders that will prevent walking,
* Having any chronic illness or psychiatric conditions or mental afflictions that may interfere with cooperation or compliance with exercise tests.

Individuals participating in the study will be informed verbally and in writing about the study protocol and informed consent form will be obtained.

ELIGIBILITY:
COVID-19 Group Inclusion Criteria

* Having been diagnosed with COVID-19 at least 12 weeks ago,
* Being literate,
* Being in the age range of 18-65,
* Volunteering to participate in research,
* To be clinically stable, to be under control if any accompanying comorbid conditions (such as hypertension, diabetes),
* Not having any orthopedic and neurological problems that might interfere with evaluating peripheral muscle strength, balance and exercise capacity.

COVID-19 Group Exclusion Criteria Those with an ICU hospitalization history due to the diagnosis of COVID-19,

* Recent myocardial infarction and pulmonary embolism.
* Having accompanying chronic diseases,
* Those who have any orthopedic or neurological disorders that will prevent walking,
* Another COVID-19 PCR Test positivity in the last 12 weeks,
* Not being able to cooperate and adapt to exercise test due to neurological influences such as cerebrovascular disease or psychiatric disorders, Healthy Group Inclusion Criteria
* Not having COVID-19,
* Being literate,
* Being in the age range of 18-65,
* Volunteering to participate in research. The Criteria for Not Including the Healthy Group in the Study
* Those who have any orthopedic or neuromuscular disorders that will prevent walking,
* Having any chronic illness or psychiatric conditions or mental afflictions that may interfere with cooperation or compliance with exercise tests.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of the study is individuals who live in Ankara and have passed the diagnosis of COVID-19 for at least 12 weeks and healthy individuals who have not had COVID-19.
  The sample of the study is healthy individuals in the long term after the diagnosis of COVID-19 at least 12 weeks after the diagnosis of COVID-19 and healthy individuals who have not had COVID-19 in Hacettepe University Adult Hospital who meet the inclusion criteria and volunteer to participate in the study.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Incremental shuttle walking test | January,2021 - December,2021
  It assesses maximal exercise capacity.

SECONDARY OUTCOMES:
Time up and Go Test | January,2021 - December,2021
  Functional balance and walking capacity
Short form McGill-Melzack Pain Questionnaire | January,2021 - December,2021
  The pain rating index has 2 subscales:
  Sensory subscale with 11 words, and Affective subscale with 4 words. These words or items are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate and 3 = severe. There's also one item for present pain intensity and one item for a 10 cm visual analogue scale (VAS) for average pain.
  The higher the total score on the MPQ, the more the pain experience for the patient increases
Tampa Kinesophobia Questionnaire | January,2021 - December,2021
  Assessment of fear of movement. Scores range from 17-68. Higher scores indicate higher level of kinesiophobia
Hospital Anxiety and Depression Scale | January,2021 - December,2021
  Assessment of anxiety and depression. Scores range from 0 to 21 for each of the two subscales. Higher scores indicate higher level of anxiety and depression
SF-36 Quality of Life Scale | January,2021 - December,2021
  Assessment of life quality. The scores of each domain ranges from zero to 100 which higher scores indicating higher levels of functioning or well-being
Fatigue Severity Scale | January,2021 - December,2021
  Assessment of fatigue perception. Scores range from 0-7. Scores higher than 4 indicate severe fatigue perception.
Cognitive Status Scale | January,2021 - December,2021
  Assessment of cognitive status. Score ranges from 0-100. Higher scores indicate increased tendency to cognitive failure.
Body Mass Index | January,2021 - December,2021
  Body mass index (BMI) is a measure of body fat based on height and weight that applies to adult men and women.
Body composition analysis with bioelectrical impedance analysis system | January,2021 - December,2021
  FM and FFM ratio

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Sain-Guven, Professor, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Barker-Davies RM, O'Sullivan O, Senaratne KPP, Baker P, Cranley M, Dharm-Datta S, Ellis H, Goodall D, Gough M, Lewis S, Norman J, Papadopoulou T, Roscoe D, Sherwood D, Turner P, Walker T, Mistlin A, Phillip R, Nicol AM, Bennett AN, Bahadur S. The Stanford Hall consensus statement for post-COVID-19 rehabilitation. Br J Sports Med. 2020 Aug;54(16):949-959. doi: 10.1136/bjsports-2020-102596. Epub 2020 May 31. PMID 32475821
- [Result] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Result] Zhao H, Shen D, Zhou H, Liu J, Chen S. Guillain-Barre syndrome associated with SARS-CoV-2 infection: causality or coincidence? Lancet Neurol. 2020 May;19(5):383-384. doi: 10.1016/S1474-4422(20)30109-5. Epub 2020 Apr 1. No abstract available. PMID 32246917
- [Result] Epidemiology Working Group for NCIP Epidemic Response, Chinese Center for Disease Control and Prevention. [The epidemiological characteristics of an outbreak of 2019 novel coronavirus diseases (COVID-19) in China]. Zhonghua Liu Xing Bing Xue Za Zhi. 2020 Feb 10;41(2):145-151. doi: 10.3760/cma.j.issn.0254-6450.2020.02.003. Chinese. PMID 32064853
- [Result] Belli S, Balbi B, Prince I, Cattaneo D, Masocco F, Zaccaria S, Bertalli L, Cattini F, Lomazzo A, Dal Negro F, Giardini M, Franssen FME, Janssen DJA, Spruit MA. Low physical functioning and impaired performance of activities of daily life in COVID-19 patients who survived hospitalisation. Eur Respir J. 2020 Oct 15;56(4):2002096. doi: 10.1183/13993003.02096-2020. Print 2020 Oct. PMID 32764112